CLINICAL TRIAL: NCT00562419
Title: Phase 2, 2-Part, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of CT-322 Monotherapy and Combination Therapy With Irinotecan in Patients With Recurrent Glioblastoma Multiforme
Brief Title: CT-322 in Treating Patients With Recurrent Glioblastoma Multiforme and Combination Therapy With Irinotecan
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adnexus, A Bristol-Myers Squibb R&D Company (Industry)
Responsible Party: Medical Director, Adnexus, A Bristol-Myers Squibb R&D Company, Adnexus, A Bristol-Myers Squibb R&D Company
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-322.002
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: Brain and Central Nervous System Tumors; Recurrent Glioblastoma Multiforme
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma | interventions — CT-322; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CT-322
  Interventions: Drug: CT-322
- 2 (Experimental): CT-322 and irinotecan hydrochloride
  Interventions: Drug: CT-322; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: CT-322 — IV solution, weekly
Drug: irinotecan hydrochloride — IV solution, biweekly
  Arms: 2

SUMMARY:
RATIONALE: CT-322 may stop the growth of glioblastoma multiforme by blocking blood flow to the tumor. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving CT-322 together with irinotecan may kill more tumor cells.

PURPOSE: This phase 2 trial is studying the side effects, tolerability, and efficacy of CT-322 when given alone and in combination with irinotecan to patients with glioblastoma multiforme.

ELIGIBILITY:
DISEASE CHARACTERISTICS

* Histologically confirmed diagnosis of recurrent/progressive GBM presenting in first, second, or third relapse (progression following anti-cancer therapy other than surgery)
* Bidimensionally measurable recurrent or residual primary disease on contrast-enhanced MRI

PATIENT CHARACTERISTICS

Age:

• 18 and over

Hematopoietic:

* ANC ≥ 1,500/mL
* Platelets ≥ 100,000/mL
* Hemoglobin ≥ 9.0g/dL

Hepatic:

* AST and ALT ≤ 1.5 x ULN
* Bilirubin ≤ 1.5 x ULN

Coagulation:

• INR < 1.5 or PT within normal limits; and PTT within normal limits

Renal:

Creatinine ≤ 1.5 x ULN; Urine protein/creatinine ratio ≤ 1

Cardiovascular

* 2-dimensional echocardiogram or cardiac multigated acquisition (MUGA) scan demonstrating left ventricular ejection fraction within the institutional normal range.
* No coronary artery bypass graft, angioplasty, vascular stenting, myocardial infarction, unstable angina, congestive heart failure within the preceding 12 months.
* No thrombotic or embolic cerebrovascular accident, including transient ischemic attacks within the past 12 months and no conditions that would not permit the safe discontinuation of specified anti-platelet medications
* No intraparenchymal CNS hemorrhage, except for Grade 1 intraparenchymal hemorrhage in the immediate post-operative period or Grade 1 intraparenchymal hemorrhage that has been stable or improved

Immunologic:

• Not known to have human immunodeficiency virus infection (HIV) or active hepatitis B or C virus infection

Other:

* Negative pregnancy test within 72 hours prior to drug administration
* Not pregnant or breast feeding
* Fertile patients must agree to use effective methods of birth control and must agree to do so until at least 4 weeks after the last dose of drug administration
* No serious non-healing wound, ulcer or bone fracture or recent significant traumatic injury (within 4 weeks)
* Have ability to understand and sign an informed consent document
* Be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* No other malignancy within the past 3 years, except for basal cell skin cancer, cervical carcinoma in situ, or other primary malignancy that is not currently clinically significant or does not require active intervention
* No prior grade 3 or greater toxicity to irinotecan
* No other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that could increase the risks associated with study participation or study drug administration or could interfere with the interpretation of the study results and would make the patient inappropriate for study entry

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 4 weeks between prior biological or immunotherapy and recovered

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered (6 weeks for nitrosoureas), unless there is unequivocal evidence of tumor progression

Radiotherapy:

• At least 12 weeks from completion of standard, daily radiotherapy and recovered, unless any of the following occurs:

* New area of enhancement on MRI that is outside the radiotherapy field
* Biopsy-proven recurrent tumor
* Radiographic evidence of progressive tumor on 2 consecutive scans taken ≥ 4 weeks apart

Surgery

* At least 4 weeks since major surgery, open biopsy or significant traumatic injury and recovered
* At least 1 week since other prior biopsy

Other:

* Not concurrently enrolled in another therapeutic clinical trial involving ongoing therapy
* No prior treatment with VEGF or VEGFR inhibitors or vascular targeting/disrupting agents
* No prior CT-322 therapy
* No prior failure of irinotecan therapy
* No prior treatment with stereotactic radiosurgery, brachytherapy, or a surgically created resection cavity to support other anatomically localized therapies
* No severe or uncontrolled medical disease (uncontrolled diabetes, hypertension, serious infection > CTCAE grade 2, significant bleeding or platelet dysfunction, gastrointestinal bleed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of CT-322 when administered alone or in combination with irinotecan hydrochloride (Part 1) | 15 ± 5 days post the last dose of study drug
Progression-free survival at 6 months (Part 2) | Measured upon initiation of cycles 2, 3, 5, 7, 9, 11, and end of study

SECONDARY OUTCOMES:
To assess the plasma pharmacokinetics of CT-322 (Cmax, Tmax, AUC, T-HALF) derived from plasma concentration vs time for CT-322 given alone and in combination with irinotecan | Part 1: cycle 1, days 1-3, day 5 or 6, days 8, 15, and 22; cycles 2-4, 6, 9, and 12, day 1; EOS and follow up visits. Part 2: cycle 1, days 1, 8, 15, and 22; cycles 2-4, 6, 9, and 12, day 1; EOS and follow up visits.
To assess the presence of anti CT-322 antibodies | Part 1: cycle 1, days 1 and 15; cycles 2-4, 6, 9, and 12, day 1; EOS and follow up visits. Part 2: cycle 1, days 1 and 15; cycles 2-4, 6, 9, and 12, day 1; EOS and follow up visits.
To assess the biological activity of CT-322 as measured by plasma biological markers and neuroimaging | Part 1: cycle 1, days 1, 2, 8, 15 and 22; cycles 2-4, 6, 9, and 12, day 1; EOS visit. Part 2: cycle 1, days 1, 8, 15 and 22; cycles 2-4, 6, 9, and 12 EOS visit.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of California, San Diego, La Jolla, California
  - University of Kentucky, Lexington, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virgina, Charlottesville, Virginia
  - University of Wisconsin Hospital, Madison, Wisconsin